CLINICAL TRIAL: NCT05897697
Title: Assessing Women's Preferences for Postpartum Thromboprophylaxis: the Prefer-Postpartum Study
Acronym: PREFER-PP
Status: Completed | Type: Observational
Sponsor: Marc Blondon (Other)
Responsible Party: Sponsor-Investigator, Marc Blondon, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: UGeneva 2021-01336
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Venous Thromboembolism; Pregnancy Related
MeSH Terms: conditions — Venous Thromboembolism | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant / postpartum women: Adult women during pregnancy or the early postpartum period (within 7 days of delivery)
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Structured interview

SUMMARY:
The preferences of pregnant women for postpartum thromboprophylaxis are largely unknown. The aims of this transversal study are to elicit the preferences of pregnant/postpartum women about postpartum thromboprophylaxis in semi-structured interviews, and to estimate the utility of the relevant health states (pulmonary embolism, deep vein thrombosis, postpartum hemorrhage, subcutaneous injections). In this second aim, the investigators will also compare the effect of 2 different techniques to estimate utilities (standard gamble vs. time trade-off), using a randomization of these techniques.

ELIGIBILITY:
Inclusion Criteria:

* women
* ongoing pregnancy or within 7 days of delivery
* fluency in French or English

Exclusion Criteria:

* fetal or neonatal death

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women in a current pregnancy or within 7 days of delivery.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Preference for postpartum thromboprophylaxis | 90 days of delivery
  Risk of postpartum venous thromboembolism at which thromboprophylaxis is preferred
Quality-of-life of pulmonary embolism, deep vein thrombosis, postpartum hemorrhage and subcutaneous injections | 90 days of delivery
  Measurements of utilities of pulmonary embolism, deep vein thrombosis, postpartum hemorrhage and subcutaneous injections, by standard gamble and time trade-off methods

CONTACTS AND LOCATIONS:
Locations (2):
- Justine Hugon-Rodin, Paris, France
- Marc Blondon, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No